CLINICAL TRIAL: NCT01487434
Title: Preventing Truancy in Urban Schools Through Provision of Social Services by Truancy Officers
Brief Title: A Randomized Study to Abate Truancy and Violence in Grades 3-9 in Chicago Public Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); U.S. Department of Education (U.S. Federal Agency); William T. Grant Foundation (Other)
Responsible Party: Principal Investigator, Jonathan Guryan, Associate Professor of Human Development and Social Policy, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00035771; R01HD067500 (NIH); R305A100706 (Other Grant/Funding Number: Institute of Education Sciences); 180140 (Other Grant/Funding Number: William T. Grant Foundation)
Record Dates: First submitted 2011-11-18; First posted 2011-12-07 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Attendance and Truancy; Student Engagement; Dropout
Keywords: Attendance; Truancy; Student engagement; Mentoring; Monitoring; Case management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Check & Connect (Experimental): Check and Connect Structured Mentoring and Case Management
  Interventions: Behavioral: Check & Connect

INTERVENTIONS:
Behavioral: Check & Connect — Structured mentoring and case management

SUMMARY:
In partnership with the Chicago Public Schools (CPS), the goal of this project is to test the effectiveness of a manualized mentoring and case management program for students in grades 1-8. Most of the current policy and research attention on dropout has focused on the dropout decision itself, even though dropout is more likely to be simply the end point of a longer-term developmental process. This project seeks to learn more about the relative effectiveness of preventing dropout through mentoring and case management programs, and to learn more about the relative effectiveness of intervening early vs. later.

DETAILED DESCRIPTION:
High school graduation is tremendously protective against involvement with crime and violence, as well as against the risk of adult poverty, unemployment, and poor health. Most of the policy and research attention on dropout has focused on the dropout decision itself. Yet dropout is almost always the end point of a longer-term developmental process. For this project the investigators have raised nearly $7 million in external support from the U.S. Department of Education, the National Institutes of Health, and the William T. Grant Foundation to learn more about the relative effectiveness of preventing dropout by trying to re-engage children in school much earlier during their academic careers.

Specifically, this project is motivated by findings from the late University of Chicago sociologist James Coleman indicating that one of the strongest protective factors against school failure for children is having a strong relationship with a pro-social adult - something that far too many children do not currently have, particularly those growing up in distressed family and community environments. The investigators are partnering with other researchers at Northwestern, Duke, and the University of Minnesota to test at large scale the effects of a structured mentoring and monitoring programs called Check & Connect. To date, the project has completed its pilot year, and starting this academic year will work with nearly 500 elementary and middle school students distributed across 23 CPS schools on the West and South sides of the city. Students will receive Check & Connect assistance for two academic years total.

ELIGIBILITY:
Inclusion Criteria:

* Student with 10-27 total absences in prior school year
* Students in Grades 1-7 at start of 2011-2012 or 2013-14 school years
* In attendance at one of the Chicago Public Schools elementary/middle schools randomly selected to be offered the intervention

Exclusion Criteria:

* None

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5300 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change in attendance and truancy | 2 times a year (on average every 6 months) during the intervention and 1 time a year each year following the completion of the intervention for up to 25 years
  Attendance and truancy measured through school records on absences

SECONDARY OUTCOMES:
Criminal activity and involvement | 1 time a year each year following the completion of the intervention for up to 25 years
  Criminal activity and involvement using criminal records will include individual-level administrative data on juvenile arrests from the Chicago Police Department and Cook County juvenile court records
Employment history and workforce involvement | 1 time a year each year following the completion of the intervention for up to 25 years
  Employment outcomes using employment records will include formal labor market involvement as measured by quarterly unemployment insurance (UI) records from the Illinois Department of Employment Security
Health and medical system participation | 1 time a year each year following the completion of the intervention for up to 25 years
  Health outcomes using health records will include Medicaid records on eligibility and service use from the Medicaid Analytic eXtract (MAX)
Academic achievement | 1 time a year each year during the intervention and 1 time a year each year following the completion of the intervention for up to 25 years
  Academic achievement measured through school records will include grades received in school and scores on standardized achievement tests (Iowa Test of Basic Skills in reading and math)
School engagement | 1 time a year each year during the intervention and 1 time a year each year following the completion of the intervention for up to 25 years
  School engagement measured through school records will include disciplinary actions/referrals

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Guryan, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Chicago Public Schools, Chicago, Illinois, United States

REFERENCES:
- [Background] Allensworth, E. M. & John Q. Easton (2007). "What Matters for Staying On-Track and Graduating in Chicago Public High Schools." Chicago, Consortium on Chicago School Research.
- [Background] Christenson, S.L, Sinclair M.F., Evelo D.L., and C.M. Hurley (1998) "Promoting school engagement with school using the Check & Connect model." Australian Journal of Guidance & Counseling, 9(1): 169-184.
- [Background] Jacob, Brian and Jens Ludwig. (2009). "Improving Educational Outcomes for Poor Children." In Changing Poverty, Changing Policies, edited by Maria Cancian and Sheldon Danziger. New York: Russell Sage Foundation.
- [Background] Sinclair, M.F., Christenson, S.L., Evelo D. L., and C.M. Hurley (1998). "Dropout prevention for youth with disabilities: Efficacy of a sustained school engagement procedure." Exceptional Children, 65(1): 7-21.
- [Background] Sinclair, M. F., Christenson, S. L. and M. L. Thurlow. (2005). "Promoting school completion of urban secondary youth with emotional and behavioral disabilities." Exceptional Children, 71(4): 465-482.
- See also: Check & Connect — http://checkandconnect.org/